CLINICAL TRIAL: NCT01265095
Title: Establish Quantitative PCR to Measure Bacteria Load of the VRE Bacteremia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201011023RB
Record Dates: First submitted 2010-12-10; First posted 2010-12-22 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Bacteremia
Keywords: VRE
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VRE bacteremia: VRE bacteremia patients

SUMMARY:
The investigators hypothesized that quantitative PCR can be used in VRE bacteremia outcome monitoring. Vancomycin-resistant enterococci (VRE) was first found in 1988 and has become an important healthcare-associated pathogen due to rapid spread, limited options for therapy and the possibility of transferring vancomycin resistance to more virulent pathogens. VRE infections not only contribute to more hospital cost and longer length of hospital stay, but also higher attributable mortality compared to those caused by vancomycin susceptible enterococci. Two different meta-analyses have shown that vancomycin resistance is an independent predictor of death among patients with enterococcal bloodstrem infections (BSIs). Despite this, few effective antibiotics are approved by the US Food and Drug Administration for the treatment of serious VRE infections. Though several studies have conducted to find the possible mortality predictors, but none has used bacterial load as a marker.

Schonheyder et al. have used semiquantitative culture, and demonstrate the relationship between high bacterial load and mortality. However, it may take more than two days before culture result available, and the sensitivity of culture is greatly affected by antimicrobial treatment. Real-time PCR has been demonstrate good performance in early detection of bacteremia, and theoretically is less affected by antimicrobial usage. However, using quantitative real-time PCR to quantify VRE in blood has not been explored, yet.

The objective of this study is to establish a quantitative method to measure the amounts of VRE in blood using the VRE specific van gene. And test the hypothesis that higher VRE load in blood results in higher mortality among patients with VRE BSIs.

Primers and probe of VRE Real-time PCR will be constructed first. The investigators will prospective enroll patient with VRE bacteremia. Clinical data and outcome will be monitored. Bacteria load of VRE bacteremia will be measured via established real-time PCR. The outcome and the association of bacteria load of VRE bacteremia will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* >18 y/o
* VRE bacteremia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: VRE bacteremia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
all cause inhospital mortality | 30days
  inhospital mortality as primary outcome, mean length of hospital stay around 30 days

SECONDARY OUTCOMES:
VRE DNA load | 14days
  VRE DNA load change during VRE treatment. Pre- and post-treatment compare.

CONTACTS AND LOCATIONS:
Overall Officials: JannTay Wang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- national Taiwan University Hospital, Taipei, Taiwan, Taiwan